CLINICAL TRIAL: NCT03209440
Title: Palliative Care for Elderly Outpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Northwestern University (Other); Rush University (Other); Emory University (Other); M.D. Anderson Cancer Center (Other); University of California, San Francisco (Other); Healthcare Chaplaincy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201601190-N; 5R01CA200867-05 (NIH); OCR17893 (Other: UF OnCore); PRO00002457 (Other: UFIRST Proposal)
Record Dates: First submitted 2017-06-26; First posted 2017-07-06 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Cancer Terminal

STUDY DESIGN:
Intervention Model Description: a 6-site, pre/posttest, randomized, controlled 4-step, stepped-wedge design to compare the effects of usual outpatient palliative care (arm 1) and usual outpatient palliative care along with nurse-led (arm 2) or chaplain-led (arm 3) DT on patient outcomes and palliative care processes. The study team will assign the 6 sites to usual care during the first-step period (approximately 12 months), and randomly assign 2 sites per step to begin and continue DT during each of the next 3 steps (12 months each).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- usual outpatient palliative care (Active Comparator): During the usual care steps, patients will receive usual outpatient palliative care
  Interventions: Behavioral: Usual care
- Dignity Therapy - Nurse Led (Experimental): During the experimental steps as part of routine palliative care service delivery, patients receive nurse-led DT.
  Interventions: Behavioral: Dignity Therapy - Nurse Led
- Dignity Therapy - Chaplain Led (Experimental): During the experimental steps as part of routine palliative care service delivery, patients will receive chaplain-led DT.
  Interventions: Behavioral: Dignity Therapy - Chaplain Led

INTERVENTIONS:
Behavioral: Dignity Therapy - Nurse Led — The nurse-led intervention involves three sessions, each of which follows a set process. The standardize approach to the delivery of the intervention facilitates a personal process of reflection and recognition that allows the patient to make meaning of their experience.
  Arms: Dignity Therapy - Nurse Led
Behavioral: Usual care — Palliative care nurses usually see patients each clinic visit to assess vital signs, function, symptoms, and to provide patient and family education. They document findings and interventions in the electronic health record (EHR). Whereas usual care for palliative care chaplaincy in the outpatient setting varies by site, chaplaincy care for usual care patients in this study will follow the usual practice for inpatient palliative care chaplaincy, which is to visit all new referrals to the clinic and assess their spiritual and religious needs. This assessment is then memorialized in a spiritual treatment plan documented in the EHR.
  Arms: usual outpatient palliative care
Behavioral: Dignity Therapy - Chaplain Led — The chaplain-led DT intervention involves three sessions, each of which follows a set process. The standardize approach to the delivery of the intervention facilitates a personal process of reflection and recognition that allows the patient to make meaning of their experience.
  Arms: Dignity Therapy - Chaplain Led

SUMMARY:
Our long-term goal is to improve spiritual care outcomes for elderly patients with cancer. The study team will use a spiritual intervention, Dignity Therapy (DT), to help these patients maintain pride, find spiritual comfort, enhance continuity of self, and ultimately make meaning of their life threatening illness.

DETAILED DESCRIPTION:
The study team propose a 3 arm pre/posttest, RCT with a 4-step (approximately 12 months per step), stepped-wedge design to compare effects of usual outpatient palliative care (usual care) and usual care along with either nurse-led or chaplain-led DT on patient outcomes, cancer prognosis awareness. The study team will assign 6 outpatient palliative care sites to usual care during the first-step, and randomly assign two sites per step to begin and continue DT led by either a nurse or a chaplain during each of the next 3 steps. During the usual care steps, 280 patients will complete pretest measures and satisfaction with palliative spiritual care services, receive usual palliative care, and complete posttest measures. During the experimental steps as part of routine palliative care service delivery, 280 patients will complete pretest measures, receive nurse-led or chaplain-led DT, and complete posttest measures. Using mixed level analysis with site, provider (nurse, chaplain) and time (step) included in the model, the study team will compare the usual care and each of the DT groups for effects on dignity impact, existential tasks, and cancer prognosis awareness and explore the moderating effects of physical symptoms and spiritual distress. The study team will also determine the effect of usual care and DT on the patient's satisfaction with palliative spiritual care services and the report of the patient's unmet spiritual needs.

ELIGIBILITY:
Inclusion Criteria:

1. cancer diagnosis (receiving cancer therapy or cancer control care)
2. receiving outpatient palliative care
3. age 55 years or older
4. able to speak and read English
5. physically able to complete the study (Palliative Performance Scale [PPS]>50, suggesting a mean in life expectancy of 53 days at the time of enrollment since each patient is expected to participate in the study for 28-42 days maximum [4-6 weeks]).

Exclusion Criteria:

1. legally blind
2. cognitively unable to complete study measures (Mini Mental Status Exam [MMSE] does not correctly spell the word world backwards)
3. history of psychosis (medical record review)
4. Patient Dignity Inventory score that indicates their distress level falls outside the remaining quota for a given step (quota is 50% of sample/site/step with low distress ≤ 2 problems rated >2 & 50% with high distress ≥ 3 problems rated >2)
5. Spiritual distress score that indicates their distress level falls outside the remaining quota for a given step (quota is 50% of sample/site/step with low distress ≤ 2 problems rated >2 & 50% with high distress ≥ 3 problems rated >2)
6. are participating in another psychosocial intervention study that is focused on concepts similar to the proposed study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana J Wilkie, PhD, Principal Investigator — University of Florida; Tammi Quest, MD, Study Director — Emory University; George Fitchett, PhD, Principal Investigator — Rush University; Michael Rabow, MD, Study Director — University of California, San Francisco; Linda Emanuel, MD/PhD, Principal Investigator — Northwestern University; Marvin Delgado, MD, Study Director — MD Anderson
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scarton LJ, Boyken L, Lucero RJ, Fitchett G, Handzo G, Emanuel L, Wilkie DJ. Effects of Dignity Therapy on Family Members: A Systematic Review. J Hosp Palliat Nurs. 2018 Dec;20(6):542-547. doi: 10.1097/NJH.0000000000000469. PMID 30379798
- [Background] Scarton L, Oh S, Sylvera A, Lamonge R, Yao Y, Chochinov H, Fitchett G, Handzo G, Emanuel L, Wilkie D. Dignity Impact as a Primary Outcome Measure for Dignity Therapy. Am J Hosp Palliat Care. 2018 Nov;35(11):1417-1420. doi: 10.1177/1049909118777987. Epub 2018 May 24. PMID 29793345
- [Background] Kittelson S, Scarton L, Barker P, Hauser J, O'Mahony S, Rabow M, Delgado Guay M, Quest TE, Emanuel L, Fitchett G, Handzo G, Yao Y, Chochinov HM, Wilkie D. Dignity Therapy Led by Nurses or Chaplains for Elderly Cancer Palliative Care Outpatients: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Apr 17;8(4):e12213. doi: 10.2196/12213. PMID 30994466
- [Result] O'Mahony S, Kittelson S, Barker PC, Delgado Guay MO, Yao Y, Handzo GF, Chochinov HM, Fitchett G, Emanuel LL, Wilkie DJ. Association of Race with End-of-Life Treatment Preferences in Older Adults with Cancer Receiving Outpatient Palliative Care. J Palliat Med. 2021 Aug;24(8):1174-1182. doi: 10.1089/jpm.2020.0542. Epub 2021 Mar 23. PMID 33760658
- [Result] Samuels V, Schoppee TM, Greenlee A, Gordon D, Jean S, Smith V, Reed T, Kittelson S, Quest T, O'Mahony S, Hauser J, Guay MOD, Rabow MW, Emanuel L, Fitchett G, Handzo G, Chochinov HM, Yao Y, Wilkie DJ. Interim Analysis of Attrition Rates in Palliative Care Study on Dignity Therapy. Am J Hosp Palliat Care. 2021 Dec;38(12):1503-1508. doi: 10.1177/1049909121994309. Epub 2021 Feb 9. PMID 33557587
- [Result] Bluck S, Mroz EL, Wilkie DJ, Emanuel L, Handzo G, Fitchett G, Chochinov HM, Bylund CL. Quality of Life for Older Cancer Patients: Relation of Psychospiritual Distress to Meaning-Making During Dignity Therapy. Am J Hosp Palliat Care. 2022 Jan;39(1):54-61. doi: 10.1177/10499091211011712. Epub 2021 Apr 29. PMID 33926243
- [Result] Schoppee TM, Scarton L, Bluck S, Yao Y, Keenan G, Handzo G, Chochinov HM, Fitchett G, Emanuel LL, Wilkie DJ. Description of a training protocol to improve research reproducibility for dignity therapy: an interview-based intervention. Palliat Support Care. 2022 Apr;20(2):178-188. doi: 10.1017/S1478951521000614. PMID 34036932
- [Result] Damen A, Exline J, Pargament K, Yao Y, Chochinov H, Emanuel L, Handzo G, Wilkie DJ, Fitchett G. Prevalence, Predictors and Correlates of Religious and Spiritual Struggles in Palliative Cancer Patients. J Pain Symptom Manage. 2021 Sep;62(3):e139-e147. doi: 10.1016/j.jpainsymman.2021.04.024. Epub 2021 May 10. PMID 33984462
- [Result] Bylund CL, Taylor G, Mroz E, Wilkie DJ, Yao Y, Emanuel L, Fitchett G, Handzo G, Chochinov HM, Bluck S. Empathic communication in dignity therapy: Feasibility of measurement and descriptive findings. Palliat Support Care. 2022 Jun;20(3):321-327. doi: 10.1017/S1478951521001188. PMID 35713352
- [Result] Rantanen P, Chochinov HM, Emanuel LL, Handzo G, Wilkie DJ, Yao Y, Fitchett G. Existential Quality of Life and Associated Factors in Cancer Patients Receiving Palliative Care. J Pain Symptom Manage. 2022 Jan;63(1):61-70. doi: 10.1016/j.jpainsymman.2021.07.016. Epub 2021 Jul 29. PMID 34332045
- [Result] Schoppee TM, Scarton L, Bluck S, Yao Y, Keenan G, Samuels V, Fitchett G, Handzo G, Chochinov HM, Emanuel LL, Wilkie DJ. Dignity therapy intervention fidelity: a cross-sectional descriptive study with older adult outpatients with cancer. BMC Palliat Care. 2022 Jan 11;21(1):8. doi: 10.1186/s12904-021-00888-y. PMID 35016670
- [Result] Handzo GF, Chochinov HM, Emanuel L, Fitchett G, Hauser J, Kittelson S, Schoppee TM, Yao Y, Solomon S, Wilkie DJ. Letter to the Editor: Feasibility of Dignity Therapy to Reduce Death Anxiety. J Palliat Med. 2022 Oct;25(10):1458-1459. doi: 10.1089/jpm.2022.0263. No abstract available. PMID 36190483
- [Result] Emanuel LL, Solomon S, Chochinov HM, Delgado Guay MO, Handzo G, Hauser J, Kittelson S, O'Mahony S, Quest TE, Rabow MW, Schoppee TM, Wilkie DJ, Yao Y, Fitchett G. Death Anxiety and Correlates in Cancer Patients Receiving Palliative Care. J Palliat Med. 2023 Feb;26(2):235-243. doi: 10.1089/jpm.2022.0052. Epub 2022 Sep 2. PMID 36067074
- [Result] Al Yacoub R, Rangel AP, Shum-Jimenez A, Greenlee A, Yao Y, Schoppee TM, Fitchett G, Handzo G, Chochinov HM, Emanuel LL, Kittelson S, Wilkie DJ. Cost considerations for implementing dignity therapy in palliative care: Insights and implications. Palliat Support Care. 2023 Aug 11:1-5. doi: 10.1017/S1478951523001177. Online ahead of print. PMID 37565429
- [Result] Wilkie DJ, Fitchett G, Yao Y, Schoppee T, Delgado Guay MO, Hauser J, Kittelson S, O'Mahony S, Rabow M, Quest T, Solomon S, Handzo G, Chochinov HM, Emanuel LL. Engaging Mortality: Effective Implementation of Dignity Therapy. J Palliat Med. 2024 Feb;27(2):176-184. doi: 10.1089/jpm.2023.0336. Epub 2023 Sep 7. PMID 37676977
- [Derived] Koch MK, Bluck S, Maggiore S, Chochinov HM, Cogdill-Richardson K, Bylund CL. Facing off-time mortality: Leaving a legacy. Psychol Aging. 2024 Jun;39(4):400-412. doi: 10.1037/pag0000815. Epub 2024 Apr 11. PMID 38602809

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: outpatient palliative care sites
Groups:
- Chaplain Sequence 1: 12 months of usual care followed by 36 months of chaplain led dignity therapy
- Nurse Sequence 1: 12 months of usual care followed by 36 months of nurse-led dignity therapy
- Chaplain Sequence 2: 24 months of usual care followed by 24 months of chaplain led dignity therapy
- Nurse Sequence 2: 24 months of usual care followed by 24 months of nurse led dignity therapy
- Chaplain Sequence 3: 36 months of usual care followed by 12 months of chaplain led dignity therapy
- Nurse Sequence 3: 36 months of usual care followed by 12 months of nurse led dignity therapy
Period: Step 1: Month 1-12
Arm/Group | Chaplain Sequence 1 | Nurse Sequence 1 | Chaplain Sequence 2 | Nurse Sequence 2 | Chaplain Sequence 3 | Nurse Sequence 3
Started | 24; 1 outpatient palliative care sites | 22; 1 outpatient palliative care sites | 28; 1 outpatient palliative care sites | 14; 1 outpatient palliative care sites | 26; 1 outpatient palliative care sites | 28; 1 outpatient palliative care sites
Completed | 22; 1 outpatient palliative care sites | 20; 1 outpatient palliative care sites | 25; 1 outpatient palliative care sites | 13; 1 outpatient palliative care sites | 25; 1 outpatient palliative care sites | 24; 1 outpatient palliative care sites
Not Completed | 2; 0 outpatient palliative care sites | 2; 0 outpatient palliative care sites | 3; 0 outpatient palliative care sites | 1; 0 outpatient palliative care sites | 1; 0 outpatient palliative care sites | 4; 0 outpatient palliative care sites
Period: Step 2: Month 13-24
Arm/Group | Chaplain Sequence 1 | Nurse Sequence 1 | Chaplain Sequence 2 | Nurse Sequence 2 | Chaplain Sequence 3 | Nurse Sequence 3
Started | 15; 1 outpatient palliative care sites (Note that the participants in each step were new participants, not those that completed the previous step.) | 11; 1 outpatient palliative care sites | 18; 1 outpatient palliative care sites | 23; 1 outpatient palliative care sites | 32; 1 outpatient palliative care sites | 20; 1 outpatient palliative care sites
Completed | 9; 1 outpatient palliative care sites | 7; 1 outpatient palliative care sites | 16; 1 outpatient palliative care sites | 23; 1 outpatient palliative care sites | 30; 1 outpatient palliative care sites | 19; 1 outpatient palliative care sites
Not Completed | 6; 0 outpatient palliative care sites | 4; 0 outpatient palliative care sites | 2; 0 outpatient palliative care sites | 0; 0 outpatient palliative care sites | 2; 0 outpatient palliative care sites | 1; 0 outpatient palliative care sites
Period: Step 3: Month 25-36
Arm/Group | Chaplain Sequence 1 | Nurse Sequence 1 | Chaplain Sequence 2 | Nurse Sequence 2 | Chaplain Sequence 3 | Nurse Sequence 3
Started | 18; 1 outpatient palliative care sites | 13; 1 outpatient palliative care sites | 24; 1 outpatient palliative care sites | 11; 1 outpatient palliative care sites | 13; 1 outpatient palliative care sites | 14; 1 outpatient palliative care sites
Completed | 11; 1 outpatient palliative care sites | 4; 1 outpatient palliative care sites | 14; 1 outpatient palliative care sites | 10; 1 outpatient palliative care sites | 12; 1 outpatient palliative care sites | 14; 1 outpatient palliative care sites
Not Completed | 7; 0 outpatient palliative care sites | 9; 0 outpatient palliative care sites | 10; 0 outpatient palliative care sites | 1; 0 outpatient palliative care sites | 1; 0 outpatient palliative care sites | 0; 0 outpatient palliative care sites
Period: Step 4: Month 37-48
Arm/Group | Chaplain Sequence 1 | Nurse Sequence 1 | Chaplain Sequence 2 | Nurse Sequence 2 | Chaplain Sequence 3 | Nurse Sequence 3
Started | 65; 1 outpatient palliative care sites | 22; 1 outpatient palliative care sites | 39; 1 outpatient palliative care sites | 44; 1 outpatient palliative care sites | 27; 1 outpatient palliative care sites | 28; 1 outpatient palliative care sites
Completed | 41; 1 outpatient palliative care sites | 9; 1 outpatient palliative care sites | 19; 1 outpatient palliative care sites | 37; 1 outpatient palliative care sites | 22; 1 outpatient palliative care sites | 24; 1 outpatient palliative care sites
Not Completed | 24; 0 outpatient palliative care sites | 13; 0 outpatient palliative care sites | 20; 0 outpatient palliative care sites | 7; 0 outpatient palliative care sites | 5; 0 outpatient palliative care sites | 4; 0 outpatient palliative care sites

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Outpatient Palliative Care | Dignity Therapy - Nurse Led | Dignity Therapy - Chaplain Led | Total
Number analyzed (Participants) | 262 | 129 | 188 | 579
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (7.5) | 65.7 (7.1) | 65.8 (7.5) | 66.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 88 | 107 | 342
  Male | 115 | 41 | 81 | 237
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 6 | 14 | 33
  Not Hispanic or Latino | 243 | 120 | 168 | 531
  Unknown or Not Reported | 6 | 3 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 68 | 21 | 14 | 103
  White | 182 | 103 | 163 | 448
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 7 | 20
Dignity Impact Scale [Mean (Standard Deviation); unit: units on a scale (7-35) higher=better] | 25.9 (4.3) | 24.3 (4.3) | 24.2 (4.2) | 25.0 (4.4)
Preparation [Mean (Standard Deviation); unit: units on a scale (4-20) higher=better] | 15.4 (3.2) | 14.5 (3.3) | 14.8 (3.7) | 15.0 (3.4)
Completion [Mean (Standard Deviation); unit: units on a scale (7-35) higher=better] | 26.8 (5.2) | 26.4 (5.9) | 27.9 (5.7) | 27.0 (5.6)
Peaceful Awareness [Count of Participants; unit: Participants]
  Peacefully aware | 59 | 32 | 40 | 131
  Not peacefully aware | 203 | 97 | 148 | 448
Treatment Preference [Count of Participants; unit: Participants]
  Prolong life; treat everything | 37 | 16 | 17 | 70
  Attempt to cure but re-evaluate often | 88 | 40 | 50 | 178
  Limit to less invasive and less burdensome interventions | 55 | 29 | 38 | 122
  Provide comfort care only | 82 | 44 | 83 | 209

OUTCOME MEASURES:

1. Primary Outcome: Dignity Impact Scale
Description: Our primary outcome measure is a 7-item Dignity Impact Scale. The items are scored on a 5-point scale from 'strongly disagree' (1) to 'strongly agree' (5). The scores can range from 7 to 35 with higher scores representing better outcome.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Outpatient Palliative Care | Dignity Therapy - Nurse Led | Dignity Therapy - Chaplain Led
Number analyzed (Participants) | 262 | 129 | 188
score on a scale | 26.3 (4.7) | 26.2 (4.1) | 26.2 (4.2)
Statistical Analysis 1: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Chaplain Led; Test type: Superiority; p = 0.02, Regression, Linear; Mean Difference (Net) = 1.67, Standard Error of Mean 0.73
Statistical Analysis 2: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Nurse Led; Test type: Superiority; p = 0.005, Regression, Linear; Mean Difference (Net) = 2.07, Standard Error of Mean 0.74

2. Secondary Outcome: Preparation
Description: Preparation for death subscale taken from the QUAL-E, a measure designed to evaluate quality of life and to assess the effectiveness of interventions targeted to improve the quality of life at the end of life. Scores range from 4 to 20 with higher scores representing better outcomes.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Outpatient Palliative Care | Dignity Therapy - Nurse Led | Dignity Therapy - Chaplain Led
Number analyzed (Participants) | 262 | 129 | 188
score on a scale | 15.6 (3.2) | 14.7 (3.2) | 14.9 (3.3)
Statistical Analysis 1: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Chaplain Led; Test type: Superiority; p = 0.21, Regression, Linear; Mean Difference (Net) = -0.62, Standard Error of Mean 0.49
Statistical Analysis 2: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Nurse Led; Test type: Superiority; p = 0.12, Regression, Linear; Median Difference (Net) = -0.79, Standard Error of Mean 0.50

3. Secondary Outcome: Completion
Description: Life completion subscale taken from the QUAL-E, a measure designed to evaluate quality of life and to assess the effectiveness of interventions targeted to improve the quality of life at the end of life. Scores range from 7 to 35 with higher scores representing better outcomes.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Outpatient Palliative Care | Dignity Therapy - Nurse Led | Dignity Therapy - Chaplain Led
Number analyzed (Participants) | 262 | 129 | 188
score on a scale | 27.0 (4.9) | 27.2 (4.9) | 28.2 (4.7)
Statistical Analysis 1: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Chaplain Led; Test type: Superiority; p = 0.21, Regression, Linear; Mean Difference (Net) = 0.90, Standard Error of Mean 0.72
Statistical Analysis 2: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Nurse Led; Test type: Superiority; p = 0.21, Regression, Linear; Mean Difference (Net) = 0.91, Standard Error of Mean 0.73

4. Secondary Outcome: Peaceful Awareness
Description: We measured peaceful awareness with the 2 items: terminal illness awareness and peaceful awareness questionnaire. The first focused on terminal illness acknowledgement (TIA) in which patients rated their current health status as 1) relatively healthy, 2) seriously but not terminally ill, or 3) seriously and terminally ill. The second item focused on the frequency of feeling deep inner peace or harmony, which was rated on a 6-point Likert scale ranging from 1) never or almost never to 6) many times a day. Scores of at least 3 on each of the two items defined positive peaceful awareness, a dichotomous measure.
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Outpatient Palliative Care | Dignity Therapy - Nurse Led | Dignity Therapy - Chaplain Led
Number analyzed (Participants) | 262 | 129 | 188
Participants
  Peacefully aware | 61 | 31 | 44
  Not peacefully aware | 201 | 98 | 144
Statistical Analysis 1: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Chaplain Led; Test type: Superiority; p = 0.11, Regression, Logistic; Odds Ratio, log = 1.00, Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Nurse Led; Test type: Superiority; p = 0.14, Regression, Logistic; Odds Ratio, log = 0.96, Standard Error of Mean 0.64

5. Secondary Outcome: Treatment Preference
Description: We measured treatment preferences with a single item from the standardized and validated Hypothetical Advanced Care Planning Scenario (H-CAP-S) that assesses treatment preferences.
Time Frame: 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Outpatient Palliative Care | Dignity Therapy - Nurse Led | Dignity Therapy - Chaplain Led
Number analyzed (Participants) | 262 | 129 | 188
Participants
  Prolong life; treat everything | 24 | 15 | 11
  Attempt to cure but re-evaluate often | 91 | 44 | 45
  Limit to less invasive and less burdensome intervention | 56 | 25 | 51
  Provide comfort care only | 91 | 45 | 81
Statistical Analysis 1: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Chaplain Led; Test type: Superiority; p = 0.05, Regression, Linear; The outcome variable was scored as 1= "prolong life; treat everything" to 4 = "provide comfort care only"; Mean Difference (Net) = 0.35, Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Usual Outpatient Palliative Care vs Dignity Therapy - Nurse Led; Test type: Superiority; p = 0.46, Regression, Linear; The outcome variable was scored as 1= "prolong life; treat everything" to 4 = "provide comfort care only"; Mean Difference (Net) = 0.13, Standard Error of Mean 0.18

ADVERSE EVENTS:
Time Frame: From baseline to posttest (about 5 weeks).
Arm/Group | Usual Outpatient Palliative Care | Dignity Therapy - Nurse Led | Dignity Therapy - Chaplain Led
All-Cause Mortality (participants affected / at risk) | 10/262 | 9/129 | 19/188
Serious Adverse Events (participants affected / at risk) | 0/262 | 0/129 | 0/188
Other Adverse Events (participants affected / at risk) | 0/262 | 0/129 | 0/188

LIMITATIONS AND CAVEATS:
Our loss to follow up was 22%, which was within our projected 20% to 30% attrition rate, but still may have unknown effects on validity of study findings. Our sample was intentionally focused on older adults with cancer. The recruited sample overrepresented the population with at least some college education and did not adequately represent the male or racial and ethnic minority populations. Future research is needed to determine the generalizability of DT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03209440/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT03209440/ICF_001.pdf